CLINICAL TRIAL: NCT04084275
Title: The Effect of Care Given Using Levine's Conservation Model on Postpartum Quality of Life in Primiparas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Şadiye Özcan, Assistant Professor Doctor, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Breastfeeding; Quality of Life; Nursing Caries; Postpartum; Nursing Model; Levine Conservation Model
Keywords: nursing care; Levine's conservation model; postpartum care; postpartum quality of life; postpartum problems
MeSH Terms: conditions — Breast Feeding | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Levine's conservation model was used as the theoretical framework for this study. A literature review was used to determine the contents of the intervention program. A nursing care program which consisted of 8 sessions, the first of which was at the hospital and the others at the homes of puerpera and which were held at different times and lasted 12 weeks in total, based on Levine's Conservation Model was provided to the women in the intervention group. Each session lasted approximately 60-120 minutes, according to the educational and practical contents.The puerpera were given trainings on different subjects based on the module during each session. For these trainings, the investigators prepared, in the light of the literature data, leaflets containing information about breastfeeding, personal hygiene, fatigue, nutrition and pilates exercises
  Interventions: Behavioral: breastfeeding education; Behavioral: personal hygiene education; Behavioral: nutrition education; Behavioral: fatigue education; Behavioral: sleep education; Behavioral: pilates exercises education
- control group (No Intervention): The puerpera in the control group received only the standard nursing care given after birth. Standard nursing care contain solely breastfeeding training. The puerpera in the control group were visited before they were discharged from the hospital to obtain their contact information and to administer them the pretest. A home visit at the end of postpartum month 3 was also planned and they were administered the posttest. After collecting the posttest data, the trainings given to the women in the intervention group on nutrition, sleep, fatigue and pilates exercises were also given to the women in the control group in consideration of the ethical dimension of the study; they were actively trained on pilates exercises by the investigator and the relevant leaflets were given to them by the end of their trainings.

INTERVENTIONS:
Behavioral: breastfeeding education
  Arms: experimental group
Behavioral: personal hygiene education — In this training, the puerpera was informed about personal hygiene to prevent infection.
  Arms: experimental group
Behavioral: nutrition education — In this training, the amount of nutrients that breastfeeding women should take daily was explained.
  Arms: experimental group
Behavioral: fatigue education — In this training, suggestions were made to prevent the negative effects of fatigue
  Arms: experimental group
Behavioral: sleep education — In this training, suggestions were offered the puerperants for better sleep. Strategies to improve sleep quality were explained.
  Arms: experimental group
Behavioral: pilates exercises education — In this study, pilates exercises exclusively for postpartum women were selected from two reference books, Fitness Professional's Handbook and Guide Women's and Fitness Health, which include 13 movements: Bridging, Hundred, Roll Up, One Leg Circle (both ways), Rocker with close legs,Single Straight Leg Stretch, Double Leg Stretch, Spine Stretch Forward, Single Leg Kick, Side Kick up and down, Side Kick circles, Rest position (stretch and relaxation) and Curling. The trainings were provided by the investigator during home visits to the puerpera in the intervention group and the pilates exercises by the investigator who was also a pilates trainer. An appropriate setting was prepared at the homes of puerpera so that they could do the pilates exercises easily.
  Arms: experimental group

SUMMARY:
Background: Postpartum period is a physiologically, emotionally and socially critical period for the woman who gave birth and also for their family. In order for women to go through their postpartum period without any problems, be able to perform self-care and have an unaffected quality of life, they need qualified, comprehensive and integrative nursing care.

Aim and objectives: This study aimed to investigate the effect of care given using Levine's conservation model on postpartum quality of life in primiparae.

Design: A randomized controlled trial. Methods: Levine's conservation model was used as the theoretical framework for this study. A literature review was used to determine the contents of the intervention program. The program consisted of 8 sessions. The puerpera were given trainings on different subjects based on the module during each session. For these trainings, the researcher prepared, in the light of the literature data, leaflets containing information about breastfeeding, personal hygiene, fatigue, nutrition and pilates exercises. The puerpera in the control group received only the standard nursing care given after birth. Standard nursing care contain solely breastfeeding training.

ELIGIBILITY:
The study included puerpera who

* were in the 18-35 age interval and were at least a primary school graduate,
* had no loss of their senses of vision or hearing,
* were open to communication and cooperation,
* had a nuclear type of family,
* were able to understand and read Turkish,
* were primiparae,
* had a full-term (between weeks 38-42) vaginal delivery,
* had a haemoglobin value of at least 10 mg/dl,
* experienced no risky conditions during gestation (placenta previa, pre-eclampsia, any systemic ailment) or during delivery (ablatio placenta, dystocia, etc.),
* were administered mediolateral episiotomy (because episiotomy impair the integrity of tissue. Healing such episiotomy incisions as soon as possible is quite important to conserve structural integrity).

Exclusion Criteria:

- those who do not meet the eligibility criteria

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed by World Health Organization Quality of Life Assessment Instrument (WHOQOL-Bref) | 3 months
  It is a multi-dimensional measurement tool designed by the World Health Organization to assess quality of life of individuals. The short form of the scale contains four domains and another domain where overall quality of life is evaluated. The domains are physical health, psychological health, social relationships, environment and general health. Each item in the scale is scored as a 5-point rating. Each domain assesses quality of life within itself independent of the others. Higher scores obtained in this scale indicate better quality of life. A study concluded that the short form of the scale was a valid and reliable instrument for the postpartum period. The validity and reliability study of the scale was performed in 1999 to be able to use it in Turkey and the Cronbach's α reliability coefficient of the scale was found to be 0.76 (Eser et al. 1999)
Fatigue assessed by Visual Analogue Scale for Fatigue | 3 months
  Developed by Lee et al. in 1991, the scale is used to measure the level of fatigue in healthy and ill individuals. Consisting of 18 items in total, the scale has 13 items to measure the level of fatigue and 5 items to measure the level of energy. There is a 10-cm horizontal line for each item of the scale with positive expressions on one end and negative on the other. Those who complete the scale are asked to mark the point which reflects best the feeling they had when they read the statement in the scale. Afterwards, the points of intersection at the places marked are measured with a ruler one by one for each question and evaluated objectively. Higher scores obtained from the fatigue items and lower scores obtained from the energy items indicate higher severity of fatigue. The validity and reliability study of the scale in Turkey and the Cronbach's α internal consistency coefficient of was found to be 0.90 (Yurtsever and Bedük, 2003).
Sleep quality assessed by Pittsburg Sleep Quality Index | 3 months
  Developed by Buysse and associates (1989), the index shows the sleep quality of an individual over the last month as stated by them. There are 19 questions in the index relating to sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction. Each question in the index is scored from 0 to 3. Zero shows having no trouble and 3 having serious trouble sleeping. Higher total scores indicate poorer sleep quality. The validity and reliability study of the index was performed in 1996 to be able to use it in Turkey and the Cronbach's α reliability coefficient of the index was found to be 0.80 (Ağargün et al.1996).

CONTACTS AND LOCATIONS:
Overall Officials: ŞADİYE ÖZCAN, Doctor, Principal Investigator — Erzincan university faculty of health sciences

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months
Access Criteria: no criteria

REFERENCES:
- [Background] Falciglia G, Piazza J, Ritcher E, Reinerman C, Lee SY. Nutrition education for postpartum women: a pilot study. J Prim Care Community Health. 2014 Oct;5(4):275-8. doi: 10.1177/2150131914528515. Epub 2014 Apr 1. PMID 24695771
- [Background] Fleming KM, Herring MP. The effects of pilates on mental health outcomes: A meta-analysis of controlled trials. Complement Ther Med. 2018 Apr;37:80-95. doi: 10.1016/j.ctim.2018.02.003. Epub 2018 Feb 13. PMID 29609943
- [Background] Gholami Z, Mohammadirizi S, Bahadoran P. Study of the Impact of Educational Behavioral Interventions on Fatigue in Mothers in the Postpartum Period in the Groups of Face-to-Face and Electronic Training. Iran J Nurs Midwifery Res. 2017 Nov-Dec;22(6):465-470. doi: 10.4103/ijnmr.IJNMR_223_15. PMID 29184586
- [Background] Hammoudeh W, Mataria A, Wick L, Giacaman R. In search of health: quality of life among postpartum Palestinian women. Expert Rev Pharmacoecon Outcomes Res. 2009 Apr;9(2):123-32. doi: 10.1586/erp.09.8. PMID 19402799
- [Background] Huang K, Tao F, Liu L, Wu X. Does delivery mode affect women's postpartum quality of life in rural China? J Clin Nurs. 2012 Jun;21(11-12):1534-43. doi: 10.1111/j.1365-2702.2011.03941.x. Epub 2011 Oct 25. PMID 22023714
- [Background] Irwin JL, Beeghly M, Rosenblum KL, Muzik M. Positive predictors of quality of life for postpartum mothers with a history of childhood maltreatment. Arch Womens Ment Health. 2016 Dec;19(6):1041-1050. doi: 10.1007/s00737-016-0653-1. Epub 2016 Aug 12. PMID 27518635
- [Background] Ko YL, Yang CL, Fang CL, Lee MY, Lin PC. Community-based postpartum exercise program. J Clin Nurs. 2013 Aug;22(15-16):2122-31. doi: 10.1111/jocn.12117. Epub 2013 Feb 9. PMID 23398359
- [Background] Phang KN, Koh SS, Chen HC. Postpartum social support of women in Singapore: A pilot study. Int J Nurs Pract. 2015 May;21 Suppl 2:99-107. doi: 10.1111/ijn.12340. PMID 26125577
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970
- [Background] Postpartum care of the mother and newborn: a practical guide. Technical Working Group, World Health Organization. Birth. 1999 Dec;26(4):255-8. PMID 10655832
- [Background] Webster J, Nicholas C, Velacott C, Cridland N, Fawcett L. Validation of the WHOQOL-BREF among women following childbirth. Aust N Z J Obstet Gynaecol. 2010 Apr;50(2):132-7. doi: 10.1111/j.1479-828X.2009.01131.x. PMID 20522068
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512